CLINICAL TRIAL: NCT00936819
Title: A Phase IIb, Randomized, Double-blind, Placebo Controlled Study Using Transplantation of Autologous Early Endothelial Progenitor Cells(EPCs) for Patients Who Have Suffered Acute Myocardial Infarction
Brief Title: The Enhanced Angiogenic Cell Therapy - Acute Myocardial Infarction Trial
Acronym: ENACT-AMI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Stem Cell Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-872; ISRCTN47943321 (Registry Identifier: controlled-trials.com)
Record Dates: First submitted 2009-07-07; First posted 2009-07-10 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anterior Wall Myocardial Infarction
Keywords: Stent; endothelial progenitor cells; nitric oxide; myocardial infarction; MRI
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Myocardial Infarction | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plasma-Lyte A and 25% autologous plasma (Placebo Comparator): A single dose of Plasma-Lyte A in Human Albumin 2.5% total = 8 mL of study product delivered into the Infarct Related Artery
  Interventions: Biological: Plasma-Lyte A and 25% Autologous Plasma
- Autologous EPCs (Experimental): A single dose of 20 million Autologous non-transfected Endothelial Progenitor Cells in Human Albumin 2.5% total = 8 mL of study product delivered into the Infarct Related Artery
  Interventions: Biological: Autologous EPCs
- Autologous EPCs Transfected with human eNOS (Experimental): A single dose of 20 million Autologous transfected with human eNOS (endothelial nitric oxide synthase) Endothelial Progenitor Cells in Human Albumin 2.5% total = 8 mL of study product delivered into the Infarct Related Artery
  Interventions: Biological: Autologous EPCs Transfected with human eNOS

INTERVENTIONS:
Biological: Plasma-Lyte A and 25% Autologous Plasma — Single dose of 8 mls given by investigator via intracoronary injection into stent of infarct-related artery
  Arms: Plasma-Lyte A and 25% autologous plasma
Biological: Autologous EPCs — Single dose of 20 million cells in 8 mls given by investigator via intracoronary injection into stent of infarct-related artery
  Other Names: Non-applicable
  Arms: Autologous EPCs
Biological: Autologous EPCs Transfected with human eNOS — Single dose of 20 million cells in 8 mls given by investigator via intracoronary injection into stent of infarct-related artery
  Other Names: Non-applicable
  Arms: Autologous EPCs Transfected with human eNOS

SUMMARY:
This will be the first clinical trial to include a strategy designed to enhance the function of autologous progenitor cells by overexpressing eNOS, and the first to use combination gene and cell therapy for the treatment of cardiac disease.

DETAILED DESCRIPTION:
Introduction:

* Despite the widespread use of pharmacological and/or interventional reperfusion therapies, recovery of cardiac function in myocardial infarction patients is often modest or in some cases absent. Unlike classical re-perfusion therapies, which must be delivered before irreversible cardiac damage has occurred, the use of progenitor cells could potentially restore functional tissue in regions that otherwise would form only scar. A number of clinical trials have been performed, mainly using autologous bone marrow cells, and these suggest a significant albeit modest improvement in cardiac function post MI. However, a major limitation of autologous cell therapy in patients with cardiovascular disease is the deleterious influence of age and other cardiac risk factors on progenitor cell activity, which may limit greatly the potential efficacy of this promising approach.

Trial Design:

* The Enhanced Angiogenic Cell Therapy - Acute Myocardial Infarction (ENACT-AMI) trial is a Canadian, 5-center, phase IIb, double-blind, parallel, randomized placebo controlled trial assessing the safety and efficacy of cell and gene therapy for patients with moderate to large anterior STEMI and who have undergone re-vascularization with stent implantation to the infarct related artery (IRA). The anticipated recruitment target is 100 patients over a two-year period.
* Consenting participants who qualify during the screening process, will undergo apheresis. Randomization, through a web-based system will take place immediately after successful apheresis. The cell collection samples will be sent to a cell manufacturing facility for manufacturing according to the treatment allocation of: a)Placebo (Plasma-Lyte A & 25% autologous plasma), b)EPCs or c)EPCs transfected with human endothelial nitric oxide synthase (eNOS).
* Approximately 5-7 days later, the patient will receive the randomized treatment allocation via intracoronary injection into the IRA. Participants will remain in hospital overnight for continuous cardiac monitoring. The first post-delivery visit will take place the following morning before hospital discharge. Subsequent study visits will be clinic visits at 1 week, 1, 3 and 6 months after study treatment. Subsequently, a registry to collect long-term safety information from telephone contacts will continue annually for 10 years. During the registry period, participants will be allowed to volunteer for enrolment in other clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-80 years of age
* Clinical diagnosis of anterior ST-elevation myocardial infarction within the last 30 days, with any one of the following 12-lead electrocardiographic changes:
* a) Greater than or equal to 1 mm ST elevation or new Q waves in 2 adjacent electrocardiographic precordial leads
* b) A new left bundle branch block AND and for patients presenting within 3 days of onset of chest pain an increase in cardiospecific enzymes (>3x CK with, EITHER positive MB fraction or increase in troponin compared to institution laboratory normal ranges)
* Successful PCI with stent implantation to infarct-related artery within the last 30 days; defined as residual stenosis no greater than 30%, TIMI flow of at least 2 or greater and a reference diameter of at least > 2mm
* Is considered hemodynamically stable at time of enrollment and immediately prior to cell delivery
* Screening LVEF must be no greater than 45% by echocardiography (determined by Simpson's method) performed at least 4 days after revascularization procedure. (All screening echos done within the first 4 days post-PCI must be repeated either by echocardiography or MRI prior to cell delivery to ensure that the variability does not exceed 10%)
* In the case of a previous myocardial infarction, documented LVEF must be 55% or greater
* Female participants MUST be surgically sterile, post-menopausal, have documented infertility, or are of child-bearing potential wih laboratory confirmation of non-pregnant state
* Provided written informed consent and is willing to comply with study follow-up visits

Exclusion Criteria:

* Significant unprotected left main disease (stenosis of 50% or greater on diagnostic angiography)
* An increase in LVEF by greater that 10% from initial LVEF evaluation for repeat assessments
* The presence of significant coronary lesions, other than the index lesion of the IRA
* A history of significant ventricular arrhythmia NOT related to index STEMI
* A history of cerebro-vascular accident or transient ischemic attack within 6 months of enrollment
* Meets at least one exclusion criterion for MRI (NB: Recent stent implantation is not an exclusion)
* Inability to undergo apheresis procedure (i.e.: poor venous access, laboratory abnormalities)
* A history of uncorrected significant valvular heart disease
* A history of left ventricular dysfunction prior to index STEMI
* A history of human immunodeficiency virus (HIV) or hepatitis B or C infection
* A history of malignancy within 5 years (Except for low-grade and fully resolved non-melanoma skin cancer)
* A history of allergy to gentamycin or amphotericin
* A history of Heparin-Induced Thrombocytopenia (HIT)
* A history of non-compliance
* Active inflammatory autoimmune disease requiring chronic immunosuppressive therapy
* Creatinine clearance <60 by Cockcroft-Gault Calculator
* Confirmed pregnant or lactating
* Is enrolled in a current investigational drug or device trial
* Participant has received cell or gene therapy in past
* The presence of any significant co-morbidities that, in the investigator's opinion, would preclude the participant from taking part in the trial
* Inability to provide informed consent and comply with the follow-up visit schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07-19 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of Global LVEF | Baseline to 6 months
  1. A change in global left ventricular ejection fraction by cardiac MRI between those treated with cell/gene enriched EPCs versus placebo
  2. Change in global left ventricular ejection fraction by cardiac MRI between those treated with non-transfected autologous EPCs versus eNOS transfected EPCs.

SECONDARY OUTCOMES:
Assessment of: Cardiac wall motion and volumes | Baseline to 6 months
  1. Change in regional wall motion and regional wall thickening by cardiac MRI between the above patient groups
  2. Change in echocardiographic assessment of LVEF, infarct size and ventricular volumes between the above patient groups
Time To Clinical Worsening (TTCW) | Baseline to 6 months
  Quality of Life Measures: Participants will complete SF-36 and DASI questionnaires at baseline, 3 and 6 months.
Safety Measurements | Baseline to 6 months
  1. Clinically significant changes in CK and troponin more than 24 hours post delivery
  2. Clinically significant changes in ECG
  3. Assessment of major acute cardiac events
  4. Evidence of any systemic embolization during the hospitalization period
  5. Need for revacularization procedures

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Stewart, MD, FRCP C, Principal Investigator — Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - L'institut de cardiologie de Montreal, Montreal, Quebec